CLINICAL TRIAL: NCT02689050
Title: Needle Based CLE in Thoracic Lymph Nodes, a Comparison With Pathology.
Brief Title: Optical Biopsy for Thoracic Lymph Nodes.
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Prof J.T. Annema, prof.dr J.T. Annema, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: NL54080.018.15
Record Dates: First submitted 2016-01-28; First posted 2016-02-23 (Estimated); Last update posted 2017-09-20 (Actual); Status verified 2017-09

CONDITIONS: Mediastinal Lymphadenopathy; Non-small Cell Lung Carcinoma; Sarcoidosis
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Sarcoidosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with lymphadenopathy: Patients ≥ 18 years of age, with (suspected) NSCLC or suspected sarcoidosis, and at least one suspected mediastinal/hilar lesion that are scheduled for standard diagnostic endosonographic workup will undergo additional needle based confocal laser endomicroscopy (nCLE) measurements of suspected lesions.
  Interventions: Device: Needle based confocal laser endomicroscopy (nCLE)

INTERVENTIONS:
Device: Needle based confocal laser endomicroscopy (nCLE) — During the fine needle aspiration of a suspected and a non-suspected lymph node we will obtain needle based CLE (nCLE) images within the lymph node. Fine needle aspirations will be obtained after the optical biopsy measurements. We will compare the results of the optical biopsy with the cytology results, or to histology in case an additional surgery is indicated.

SUMMARY:
EUS-FNA is the recommended diagnostic examination of choice when patients present with suspected lower mediastinal lymph nodes on imaging. EUS-FNA is minimal invasive and low in costs, and although it has a good record in detecting diseases (eg confirm a nodal metastasis or granulomas) it has limitations in excluding diseases (missing metastases/ or granulomas) resulting in a false negative rate of 15-20%. Substantial limitations that most likely can be attributed to areas within the node that are not sampled during EUS-FNA tissue acquisition. Improved needle based EBUS/ EUS guided nodal diagnostics might result in improved quality of the fine needle aspirations, reduce in surgical diagnostic procedures , reduced costs and result in a shorter timebefore-treatment interval.

DETAILED DESCRIPTION:
Needle based confocal laser endomicroscopy (nCLE) is a modern imaging technique, compatible with the conventional diagnostic aspiration needle, that uses an excitation laser light to create 'real-time' microscopic images of tissues. Therefore this technique provides additional information regarding the nodal status and could therefore improve the diagnostic yield of EUS-FNA. Specifically, we will describe the nCLE image characteristics of lymph nodes involved in lung cancer and sarcoidosis as well as in healthy lymph nodes. Improved characterization of mediastinal nodes might lead to improved diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Suspected or tissue proven sarcoidosis (stage I or II based on CT/PET-CT) and referred for diagnostic endosonographic work up or
* Suspected or tissue proven NSCLC with suspected mediastinal lymph nodes within reach of EUS-FNA

Exclusion Criteria:

* Inability and willingness to provide informed consent
* Inability to comply with the study protocol
* Patients with known allergy for fluorescein
* use of betablokker within 24 hours before procedure
* possible pregnancy or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with suspected non-small cell lungcarcinoma/sarcoidosis scheduled for EUS-FNA.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-01-13 (Actual); Primary Completion 2017-03-22 (Actual); Study Completion 2017-03-22 (Actual)

PRIMARY OUTCOMES:
The differences on CLE imaging between different disease entities in thoracic lymph nodes (e.g. malignant, reactive and nodes involved in sarcoidosis). | cross-sectional (2 weeks)
  follow up of 2 weeks after measurements

SECONDARY OUTCOMES:
Creating a CLE-image atlas for reactive lymph nodes and lymph nodes involved in lung cancer and sarcoidosis. | cross sectional (2 weeks)
The number of participants with procedure related adverse advents. | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jouke T Annema, MD, PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC)
Locations (1):
- Academisch Medisch Centrum, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to share nCLE results

REFERENCES:
- [Derived] Kramer T, Wijmans L, van Heumen S, Bansal S, Jeannerat D, Manley C, de Bruin M, Bonta PI, Annema JT. Needle-based confocal laser endomicroscopy for real-time granuloma detection. Respirology. 2023 Oct;28(10):934-941. doi: 10.1111/resp.14542. Epub 2023 Aug 10. PMID 37562791
- [Derived] Wijmans L, Baas P, Sieburgh TE, de Bruin DM, Ghuijs PM, van de Vijver MJ, Bonta PI, Annema JT. Confocal Laser Endomicroscopy as a Guidance Tool for Pleural Biopsies in Malignant Pleural Mesothelioma. Chest. 2019 Oct;156(4):754-763. doi: 10.1016/j.chest.2019.04.090. Epub 2019 May 7. PMID 31075217